CLINICAL TRIAL: NCT05435326
Title: The Relationship of Stump Length With Muscle Strength, Balance, and Proprioception in Patients With Traumatic Unilateral Transfemoral Amputation
Brief Title: The Relationship of Stump Length With Muscle Strength in Patients With Traumatic Unilateral Transfemoral Amputation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Associate professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 28
Record Dates: First submitted 2022-06-23; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Amputation, Traumatic
Keywords: amputation; stump length; muscle strength; balance; proprioception
MeSH Terms: conditions — Amputation, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Amputation is the loss or removal of a body part such as an arm or leg. It is the last option in trauma treatment and irreversible procedure. Amputation rehabilitation begins in the pre-amputation period. The goal of rehabilitation after an amputation is to help the patient return to the highest level of function and independence possible, while improving the overall quality of life. Many factors can affect the success of lower limb amputation rehabilitation, and stump length is one of them. A sufficient stump length provides a large contact surface and increases the stability of the socket unit.

DETAILED DESCRIPTION:
Amputation is the loss or removal of a body part such as an arm or leg. It is the last option in trauma treatment and irreversible procedure. Amputation rehabilitation begins in the pre-amputation period. The goal of rehabilitation after an amputation is to help the patient return to the highest level of function and independence possible, while improving the overall quality of life. Many factors can affect the success of lower limb amputation rehabilitation, and stump length is one of them. A sufficient stump length provides a large contact surface and increases the stability of the socket unit.

People with unilateral transfemoral amputation have lost their knee and ankle joint.

This causes a loss of proprioceptive feedback from the ankle joint, knee joint and related muscles. Muscle weakness, muscle atrophy and balance problems are common in amputee patients.

There is not enough data to reveal the relationship between stump length and muscle strength, balance, and proprioception. The aim of this study to evaluate the relationship of stump length with muscle strength, balance, and proprioception in patients with traumatic unilateral transfemoral amputation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* Time after amputation ≥ 6 months
* Unilateral transfemoral traumatic amputation

Exclusion Criteria:

* Bilateral transfemoral amputation
* Unilateral non-traumatic transfemoral amputation
* Presence of neurological, auditory, or vision-related disease that may affect balance and proprioception
* Presence of cardiovascular or pulmonary disease that will affect muscle strength

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-65 who underwent traumatic amputation at least 6 months ago will participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2022-07-18 (Estimated); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
The isokinetic muscle strength of the hip extensors and flexors | through study completion, an average of one month
  The isokinetic muscle strength of the hip extensors and flexors will be measured with the computer -assisted isokinetic system (CYBEX). The tests were performed at the angular velocities of 60° and 120°/s, while measuring flexion and extension of the amputated side.

SECONDARY OUTCOMES:
The Berg Balance Scale (BBS) | through study completion, an average of one month
  The balance will be evaluated using the Berg Balance Scale (BBS). The BBS is a clinical test commonly used to assess the patients' static and dynamic balance performance. Berg Balance Scale consist of 14 items. A participant's performance on each task is graded using a 5-point ordinal scale ranging from 0 to 4. Total score of scale is 0-56 points. The higher the scores show the better the balance ability of the patients.
Proprioception assessment | through study completion, an average of one month
  The computer-assisted isokinetic system (CYBEX) will be also used to evaluate the lower extremity proprioceptive sense of patients. The average proprioceptive errors at 15-45° and 30-60° were assessed. Patients will be taught the initial 15° and the targeted 45° hip flexion angles by keeping hip in these angles for 10 seconds. Afterwards, patients will be asked to move from the initial 15° to the target 45° while their eyes are closed. The average proprioceptive errors which are deviations from target angles will be noted. The same procedure will be done for initial 30° and target 60° angles.

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Kılınç Kamacı, MD, Principal Investigator — Specialist

REFERENCES:
- [Derived] Kilinc Kamaci G, Orucu Atar M, Ozcan F, Demir Y, Aydemir K. Relationship of stump length with muscle strength, proprioception, and balance in patients with traumatic unilateral transfemoral amputation. Prosthet Orthot Int. 2024 Dec 18;49(3):268-273. doi: 10.1097/PXR.0000000000000385. PMID 39692742